CLINICAL TRIAL: NCT00453453
Title: BNP Therapy Observation Unit Outcomes STudy
Brief Title: BNP Therapy Observation Unit Outcomes STudy (BOOST)
Acronym: BOOST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas Ander MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00038961; 0009-2006 (Other: Other)
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure; observation unit; nesiritide
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nesiritide (Experimental): Subjects who come into the ED with CHF will be treated with nesiritide
  Interventions: Drug: Nesiritide
- Standard care (No Intervention): Subjects who come into the ED with CHF will receive standard care treatment

INTERVENTIONS:
Drug: Nesiritide — Nesiritide given orally in the emergency department
  Other Names: Natrecor
  Arms: Nesiritide

SUMMARY:
The investigators hypothesize that patients admitted to an emergency department (ED) observation unit will have a decreased rate of hospital admissions and ED recidivism when treated with nesiritide versus standard therapy. The investigators also hypothesize that decreasing B-type Natriuretic Peptide (BNP) levels during treatment in an ED observation unit will predict improved patient outcomes.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a growing problem in the United States. The increasing number of decompensated heart failure patients presenting to emergency departments (ED) for treatment is worsening the burden on already strained and limited health care resources. In addition, many of these patients will return to the ED for treatment within three months of being treated for decompensated heart failure. The emergence of ED observation units has provided a viable and cost effective alternative to inpatient treatment for many diseases including CHF. It has been shown that intensive, directed therapy in ED observation units has decreased the revisit rates for CHF patients. In addition, the introduction of nesiritide has shown promising results in the treatment of decompensated congestive heart failure.

The primary aim of this study is to compare nesiritide versus standard heart failure therapy in an ED setting. A secondary aim is to determine if serial BNP levels during this observation unit stay will predict clinical outcomes.

The treatment of heart failure in the ED places a tremendous burden on already limited resources. The costs of treatment as well as the morbidity and mortality associated with the disease are worsening and are predicted to increase as the general population ages. The ability to safely treat and discharge patients from an ED observation unit while reducing return visits would be invaluable in managing the growing number of heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 years of age
* Have a working diagnosis of HF, as determined by the emergency physician using the Boston Criteria. A score of 8-12 is required for inclusion in the study.
* Alert, oriented and able to provide informed consent.
* Able to be contacted by telephone for follow up after discharge, and have none of the study exclusion criteria.

Exclusion Criteria:

* Dialysis Dependent Renal Failure
* Temperature > 38.5 degrees celsius
* Pneumonia (Infiltrates on Chest X-ray)
* Requiring IV vasoactive agents (Other than Nesiritide)
* Killip Class III/IV
* Systolic blood pressure < 90 mmHg
* EKG diagnostic or suggestive of Acute myocardial infarction or ischemia
* Abnormal Cardiac Markers
* Lack of a telephone
* Inability to provide informed consent due to cognitive impairment or a severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects that return to the emergency department in 90 days | 90 days

SECONDARY OUTCOMES:
Correlation between BNP levels at admission and number of subjects who return to the emergency department | 90 days
  The BNP levels per subject will be plotted to their return rate to the emergency department. Pearson correlation coefficient will be calculated to explore their relationship. Pearson correlation coefficient is a measure of the linear correlation (dependence) between 2 variables, giving a value between +1 and -1 inclusive, where 1 is total positive correlation, 0 is no correlation, and -1 is total negative correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ander, MD, Principal Investigator — Emory University; Daniel Wu, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hosptial, Atlanta, Georgia, United States